CLINICAL TRIAL: NCT04154540
Title: Study of Gait and Posture in Subacute Acquired Neuropathies and in Hereditary Neuropathies
Brief Title: Posturography-Neuropathy
Acronym: PONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_17; 2017-A02861-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-08-14; First posted 2019-11-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Neuropathy Demyelinating
Keywords: Gait; Balance; Posture; Charcot-Marie-Tooth; Chronic inflammatory demyelinating polyneuropathy
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- demyelinating hereditary neuropathy (Experimental): adult patients with demyelinating hereditary neuropathy type CMT 1A.
  Interventions: Other: Motion analysis
- demyelinating inflammatory neuropathy (Experimental): adult patients with acquired demyelinating inflammatory neuropathy.
  Interventions: Other: Motion analysis

INTERVENTIONS:
Other: Motion analysis — Gait and posture recording

SUMMARY:
If the classification between hereditary and acquired neuropathy is often easy, there is no completely specific marker allowing the distinction between the two etiologies. Clinical experience suggests that hereditary neuropathies have less impact on balance and gait than the acquired neuropathies at equivalent level of impairment, but this has never been clearly demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* CMT1A for molecular-proven Group 1 (PMP22 duplication)
* IPDC likely or defined for Group 2
* Able to walk 10 m unassisted

Exclusion Criteria:

* Neurological history other than neuropathy: epilepsy, stroke, dementia
* Pregnant women
* Person under guardianship or trusteeship
* Musculoskeletal conditions other than neuropathy impairing walking abilities
* Major comorbidity considered a contraindication by the investigator (cancer, unstable angor, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Posturography (Romberg's quotient) | Time 0 ; single session

SECONDARY OUTCOMES:
The Timed Up and Go test (TUG) | Time 0 ; single session
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
  the scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls
stride length (in millimeters) parameters | Time 0 ; single session
  Kinematic and Kinetic parameters of the gait initiation and the stabilised gait using the optoelectronic system (VICON®)
stride time (in seconde) parameters | Time 0 ; single session
  Kinematic and Kinetic parameters of the gait initiation and the stabilised gait using the optoelectronic system (VICON®)
velocity (meter/seconde) parameters | Time 0 ; single session
  Kinematic and Kinetic parameters of the gait initiation and the stabilised gait using the optoelectronic system (VICON®)
cadence (step/min) parameters | Time 0 ; single session
  Kinematic and Kinetic parameters of the gait initiation and the stabilised gait using the optoelectronic system (VICON®)

CONTACTS AND LOCATIONS:
Overall Officials: Céline TARD, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

REFERENCES:
- [Result] Dupont L, Defebvre L, Davion JB, Delval A, Tard C. Postural balance and visual dependence in patients with demyelinating neuropathies differ between acquired and hereditary etiologies. Rev Neurol (Paris). 2025 Jan-Feb;181(1-2):98-105. doi: 10.1016/j.neurol.2024.10.002. Epub 2024 Oct 28. PMID 39462724